CLINICAL TRIAL: NCT05409612
Title: Multicenter, Randomized, Open, Phase III, Trial Assessing the Immunogenicity and Safety of Two Influenza Vaccine Strategies Among Severe Obese Adult Patients
Brief Title: Trial Assessing the Immunogenicity and Safety of Two Influenza Vaccine Strategies Among Severe Obese Adult Patients
Acronym: FLUO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Sanofi Pasteur, a Sanofi Company (Industry); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP200039; 2021-002691-39 (EudraCT Number)
Record Dates: First submitted 2022-05-20; First posted 2022-06-08 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-01

CONDITIONS: Morbid Obesity; Severe Obesity
Keywords: Obesity; influenza vaccine; immunological response; RIV4
MeSH Terms: conditions — Obesity, Morbid; Obesity; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supemtek® arm (Active Comparator): Patients recieving a quadrivalent recombinant high-dose influenza vaccine containing 45 µg of hemagglutinin (HA) for each of the 4 strains included (2 strains A and 2 strains B).
  Solution for injection is sterile liquid supplied in 0.5mL single dose pre-filled syringe. Vaccine is injected intra-muscularly in the non-dominant arm at Day 0.
  Interventions: Biological: Supemtek®
- Vaxigriptetra® arm (Active Comparator): Patients receiving a quadrivalent inactivated influenza vaccine containing 15 µg of hemagglutinin (HA) for each of the 4 strains included. Suspension for injection is sterile liquid supplied in 0.5mL single dose pre-filled syringe. Vaccine is injected intra-muscularly in the non-dominant arm at Day 0.
  Interventions: Biological: Vaxigriptetra®

INTERVENTIONS:
Biological: Supemtek® — Quadrivalent recombinant high-dose influenza vaccine containing 45 µg of hemagglutinin (HA) for each of the 4 strains included (2 strains A and 2 strains B).
  Solution for injection is sterile liquid supplied in 0.5mL single dose pre-filled syringe. Vaccine is injected intra-muscularly in the non-dominant arm at Day 0.
  Arms: Supemtek® arm
Biological: Vaxigriptetra® — Quadrivalent inactivated influenza vaccine containing 15 µg of hemagglutinin (HA) for each of the 4 strains included. Suspension for injection is sterile liquid supplied in 0.5mL single dose pre-filled syringe. Vaccine is injected intra-muscularly in the non-dominant arm at Day 0.
  Arms: Vaxigriptetra® arm

SUMMARY:
Obesity has been considered as a risk factor for mortality and development of complications during infection with the influenza virus. Several case studies of severe and fatal infections have identified possible effects of obesity on disease progression; these effects include extensive viral replication in the deep lung, progression to viral pneumonia, and prolonged and increased viral shedding. These points may be linked to obesity which causes a chronic state of meta-inflammation with systemic implications for immunity: obese patients exhibit delayed and blunted innate and adaptive immune responses to influenza virus infection, and they experience poor recovery from the disease leading to an increased susceptibility to secondary bacterial infections and poor healing of the lung epithelium. Furthermore, in obese people, influenza virus may exploit the lack of antiviral pressure, generate a more virulent population and increase disease severity Due to the growing prevalence of obesity worldwide (500 million subjects in 2017), it is important to be able to offer vaccines that provide the highest protection for this at-risk population. The quadrivalent recombinant high-dose influenza vaccine has been shown to have greater immunogenicity and efficacy than standard influenza vaccine in non-obese adults older than 50 years. However, this vaccine has never been evaluated in obese subjects.

Investigators thus planned this trial to assess whether the use of the new quadrivalent recombinant high-dose influenza vaccine (RIV4) will induce a better immunological answer than current quadrivalent standard vaccine (SD) in patients with severe obesity, with an acceptable safety profile, thus leading to a better protection against influenza in this population at high risk of influenza complications.

DETAILED DESCRIPTION:
Obese adults are at higher risk of complications and mortality due to influenza infections than healthy adults. The few studies available showed lower vaccine response in obese patients compared to healthy adults and moderate efficacy of standard influenza vaccines among these subjects.

Data from the population > 50 years show that a recombinant high dose quadrivalent vaccination strategy improve immunological and clinical efficacy against influenza with comparable rates of local and general solicited reactions.

Investigators hypothesize that the use of the new quadrivalent recombinant high-dose influenza vaccine (RIV4) will induce a better immunological answer than current quadrivalent standard vaccine (SD) in patients with severe obesity, with an acceptable safety profile, thus leading to a better protection against influenza in this population at high risk of influenza complications.

The primary objective is to assess if the immune response of the new quadrivalent recombinant high-dose influenza vaccine (RIV4) is superior to the current quadrivalent standard dose influenza vaccine (SD) in adult patients with severe obesity in terms of geometric mean titers (GMTs) for each strain at 1 month. The primary endpoint: Ratio (RIV4/SD) of GMTs of each of the 4 strains at 1-month post-vaccination. The ratio of GMTs will be computed by taking the antilog of the difference between means of log-transformed titers.

It is a Randomized, open, multicenter, trial in France, evaluating the immunological response and safety of two influenza vaccine strategies using a standard quadrivalent vaccine (Vaxigriptetra®) and the new high-dose recombinant quadrivalent vaccine (Supemtek®). The single administration of influenza vaccine will be performed at D0: Vaxigriptetra® or Supemtek® according to randomization allocation. Three follow-up visits will be performed at M1 and M6 during consultations in the clinical units where participants are usually followed. This multicenter research will involve the participation of the 10 centers in France (metropolitan France and French overseas departments and territories). Each hospital involves a single participating department. All investigational sites belong to the FORCE (national network of clinical research specializing in the study of obesity and associated metabolic diseases) or to the I-REIVAC (Innovative Clinical Research Network In Vaccinology). The duration of recruitment will be 5 months. The duration of participation for each participant will be 6 months, the total duration of the study will be 11 months. For this study, 206 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 and ≤75 years old
2. Body Mass Index (BMI) ≥35 kg/m2
3. No previous vaccination against influenza (in the preceding 6 months) with either the trial vaccine or another vaccine
4. Absence of health event satisfying the definition of a serious adverse event, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within 15 days prior to enrolment.
5. Signed informed consent
6. Participants covered by social security regimen .

Exclusion Criteria:

1. Known active infection with HIV and / or HBV (HBs antigen) and / or HCV (RNA positive viral load)
2. Immunodepression or diagnosis of having congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus, rheumatoid arthritis, juvenile rheumatoid arthritis, inflammatory, bowel disease, or other autoimmune condition
3. Known acute evolving neurological disorder or history of Guillain-Barré syndrome.
4. Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (tympanic temperature ≥38°C on the day of vaccination). A subject should not be included in the trial until the condition has resolved or the febrile event has subsided.
5. Proven Influenza infection in the 6 months preceding the study
6. Known systemic hypersensitivity to any of the vaccine components, including a documented allergy to egg proteins, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances.
7. Receipt of any vaccine in the 2 weeks (14 days) preceding the trial vaccination
8. History of bariatric surgery in the 2 years preceding the study.
9. Bariatric surgery planned during the study period.
10. Receipt of immune globulins, blood or blood-derived products in the 3 months preceding the study or planned during the study period.
11. Taking immunosuppressive treatment (including chemotherapy, oral corticosteroids with doses ≥10 mg/day of prednisone or equivalent during ≥15 days) or radiotherapy in the 6 months preceding the study or planned during the study.
12. Contraindication to intramuscular injection
13. Female subjects of childbearing potential :

    * without an adequate contraception (see chapter 5.8) for 30 days prior to vaccination within the context of the study,
    * breastfeeding
    * with a positive pregnancy test on the day of vaccination,
    * did not agreed to continue adequate contraception during 2 months after completion of the vaccination.
14. Participation at the time of trial enrollment (or in the 4 weeks [28 days] preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
15. Anticipated inability to follow the protocol requirements (e.g. comprehension of the study requirements, ability to comprehend and comply with procedures for collection of safety data, expressed availability for the required study period, and ability and willingness to attend scheduled visits). 16. Participants covered by AME.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Ratio (RIV4/SD) of geometric mean titers (GMTs) of each of the 4 strains at 1-month post-vaccination.obesity in terms of geometric mean titers (GMTs) for each strain at 1 month. | 1 month
  The ratio of GMTs will be computed by taking the antilog of the difference between means of log-transformed titers.

SECONDARY OUTCOMES:
seroconversion rate for each of the 4 strains at 1 month after vaccination | 1 month
  defined as pre-vaccination hemagglutination inhibition (HI) titer of <1:10 and post-vaccination titer ≥1:40 or pre-vaccination HI titer of ≥ 1:10 and a 4-fold post-vaccination rise in antibody titer. Pre-vaccination titers are measured at inclusion and post-vaccination titers at 1 and 6 months after vaccination.
seroconversion rate for each of the 4 strains at 6 month after vaccination | 6 month
  (defined as pre-vaccination hemagglutination inhibition (HI) titer of <1:10 and post-vaccination titer ≥1:40 or pre-vaccination HI titer of ≥ 1:10 and a 4-fold post-vaccination rise in antibody titer. Pre-vaccination titers are measured at inclusion and post-vaccination titers at 1 and 6 months after vaccination).
seroconversion factor (or geometric mean fold increase) for each of the 4 strains at 1 month after vaccination. | 1 month
  defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the day 0 reciprocal HI titer
seroconversion factor (or geometric mean fold increase) for each of the 4 strains at 6 month after vaccination. | 6 month
  defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the day 0 reciprocal HI titer
seroprotection rate defined as the post-vaccination HI titer ≥1:40 for each of the 4 strains at 1 month after vaccination. | 1 month
  seroprotection rate defined as the post-vaccination HI titer ≥1:40 for each of the 4 strains at 1 month after vaccination.
seroprotection rate defined as the post-vaccination HI titer ≥1:40 for each of the 4 strains at 6 month after vaccination. | 6 month
  seroprotection rate defined as the post-vaccination HI titer ≥1:40 for each of the 4 strains at 6 month after vaccination.
geometric means titers at 6 months after vaccination for each of the 4 strains. | 6 month
  geometric means titers at 6 months after vaccination for each of the 4 strains.
Seroconversion rate of geometric mean titers (GMTs) of each of the 4 strains at 1 month after vaccination according to class of age (< or ≥ 50 years old) and BMI class ([35-40[ or ≥ 40 kg/m2). | 1 month
  The ratio of GMTs will be computed by taking the antilog of the difference between means of log-transformed titers
Seroconversion rate of geometric mean titers (GMTs) of each of the 4 strains at 6 month after vaccination according to class of age (< or ≥ 50 years old) and BMI class ([35-40[ or ≥ 40 kg/m2). | 6 month
  The ratio of GMTs will be computed by taking the antilog of the difference between means of log-transformed titers
seroconversion factor of geometric mean titers (GMTs) of each of the 4 strains at 1 month after vaccination according to class of age (< or ≥ 50 years old) and BMI class ([35-40[ or ≥ 40 kg/m2). | 1 month
  The ratio of GMTs will be computed by taking the antilog of the difference between means of log-transformed titers
seroconversion factor of geometric mean titers (GMTs) of each of the 4 strains at 6 month after vaccination according to class of age (< or ≥ 50 years old) and BMI class ([35-40[ or ≥ 40 kg/m2). | 6 month
  The ratio of GMTs will be computed by taking the antilog of the difference between means of log-transformed titers
seroprotection rate of geometric mean titers (GMTs) of each of the 4 strains at 1 month after vaccination according to class of age (< or ≥ 50 years old) and BMI class ([35-40[ or ≥ 40 kg/m2). | 1 month
  The ratio of GMTs will be computed by taking the antilog of the difference between means of log-transformed titers
seroprotection rate of geometric mean titers (GMTs) of each of the 4 strains at 6 month after vaccination according to class of age (< or ≥ 50 years old) and BMI class ([35-40[ or ≥ 40 kg/m2). | 6 month
  The ratio of GMTs will be computed by taking the antilog of the difference between means of log-transformed titers
ratio (RIV4/SD) of geometric mean titers (GMTs) of each of the 4 strains at 1 month after vaccination according to class of age (< or ≥ 50 years old) and BMI class ([35-40[ or ≥ 40 kg/m2). | 1 month
  The ratio of GMTs will be computed by taking the antilog of the difference between means of log-transformed titers
ratio (RIV4/SD) of geometric mean titers (GMTs) of each of the 4 strains at 6 month after vaccination according to class of age (< or ≥ 50 years old) and BMI class ([35-40[ or ≥ 40 kg/m2). | 6 month
  The ratio of GMTs will be computed by taking the antilog of the difference between means of log-transformed titers
Number and intensity of solicited reactogenicity events, clinical events within 7 days of vaccination and all other unsolicited adverse event during the study. | 1 and 6 months
  reactogenicity events : local (pain, tenderness, induration, redness, swelling) and general (tiredness, chills, joint pain, muscle pain, headache, nausea, fever)
Identification of the influenza vaccine response determinants in terms of seroconversion for at least two strains after vaccination | 1 and 6 months
  considering age, sex, smoking, BMI, chronic conditions (e.g. diabetes mellitus), co-treatments, standard / recombinant vaccine
Proven influenza cases during the study period. | 1 and 6 months
  A proven influenza infection will be defined as a positive influenza RT-PCR performed on a naso-pharyngeal swab at the time of the visit.

CONTACTS AND LOCATIONS:
Overall Officials: Odile LAUNAY, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitie-Salpêtrière hospital APHP, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodological sound proposal.